CLINICAL TRIAL: NCT04011280
Title: Novel Pharmacotherapy Approaches in Smokers With Serious Mental Illness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Veterans Medical Research Foundation (Other); University of California (Other)
Responsible Party: Principal Investigator, Robert Anthenelli, MD, Principal Investigator and Study Physician, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 180785
Record Dates: First submitted 2019-06-25; First posted 2019-07-08 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Bipolar Disorder; Schizophrenia; Schizoaffective Disorder; Nicotine Dependence
Keywords: nicotine; varenicline; Acceptance and Commitment Therapy; schizophrenia; schizoaffective; bipolar; smoking cessation; cigarette
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia; Psychotic Disorders; Tobacco Use Disorder; Smoking Cessation | interventions — Varenicline; Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: This pilot trial is a Phase IV, 12-week, single center, randomized, double blind, parallel group comparison of low (0.5 mg twice daily with slower titration over one full week) versus standard dose (1.0 mg twice daily with standard titration) varenicline in individuals with DSM-V BD or SSD with a 12-week, post-treatment follow-up.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Everyone, with the exception of the study pharmacist, will be blinded to which arm participants will be randomized into.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Low Dose Varenicline (Experimental): 0.5 mg twice daily with 0.5 mg daily titration over one full week
  Interventions: Drug: Varenicline
- Standard Dose Varenicline (Active Comparator): 1.0 mg twice daily with standard titration
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — The ten 30-minute sessions will target core processes in ACT such as acceptance and being present.
  Other Names: Acceptance and Commitment Therapy

SUMMARY:
Approximately 60 chronic smokers with bipolar disorder, schizophrenia or schizoaffective disorder who are motivated to try to quit smoking will be randomized to receive smoking cessation treatment with the FDA-approved medication, varenicline, delivered either a) at its standard dose and titration schedule (half of the participants) versus b) at a lower dose and slower titration schedule (the other half), for 12 weeks. All smokers will choose a target quit date sometime between 8 to 35 days after starting the medication. All participants will receive ten 30-minute sessions of a behavioral treatment called Acceptance and Commitment Therapy (ACT). Participants will be followed for an additional 12 weeks off study medication. The major endpoint is the feasibility of combining ACT with the different dosing strategies. Investigators will also conduct a blood test that measures the breakdown of nicotine in the body to explore whether that measure influences treatment response and side effects.

DETAILED DESCRIPTION:
This pilot feasibility trial is a Phase IV, 12-week, single center, randomized, double blind, parallel group comparison of low (0.5 mg twice daily with slower titration over one full week) versus standard dose (1.0 mg twice daily with standard titration) varenicline in individuals with DSM-V Bipolar Disorder (BD) or Schizophrenia Spectrum Disorders (SSD) with a 12-week, post-treatment follow-up. The 16 visits after screening (Weeks 0-24) include 11 in-person (with medications dispensed at weeks 0, 2, 4, 6, 8 and 10] and 5 via telephone. Plasma will be obtained at baseline to measure participants' Nicotine Metabolite Ratio (NMR) and to identify slow versus normal nicotine metabolisers. A flexible quit date (between days 8-35) will be employed allowing varenicline preloading to occur prior to the Target Quit Date. Ten sessions of Acceptance & Commitment Therapy (ACT) for smoking cessation will be delivered by trained counselors.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age
* Outpatients with a DSM-V diagnosis of Bipolar Disorder or Schizophrenia Spectrum Disorder
* Smoke at least 10 cigarettes per day and have an expired carbon monoxide (CO) breathalyzer of ≥ 10 ppm at screening and baseline visits
* Are motivated to quit smoking
* Have access to a mental health provider

Exclusion Criteria:

* Females who are pregnant, planning to become pregnant, or lactating
* Test positive for any non-prescribed medications or illicit drugs
* Have made a suicide attempt or engaged in self-mutilatory behavior in the past year
* Meet criteria for another Substance Use Disorder in the past month
* In the investigators' judgement, are either psychiatrically or medically unstable to safely participate
* Are currently using any other form of treatment for smoking cessation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pacific Treatment & Research Center at UCSD, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol defined all participants who signed a written informed consent and who completed a formal screening process as "Enrolled" in the trial. Thus, following CONSORT diagram terminology, there were N = 39 enrollees. 28 participants were randomized into one of the two treatment arms and were thus allocated to treatment.
Period: Overall Study
Arm/Group | Low Dose Varenicline | Standard Dose Varenicline
Started | 14 | 14
Completed | 9 | 12
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Varenicline | Standard Dose Varenicline | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (9.8) | 45.6 (11.6) | 47.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 13 | 13 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 8 | 6 | 14
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 14 | 28
Diagnosis: Bipolar Disorder (BD) or Schizophrenia Spectrum Disorder (SSD) [Count of Participants; unit: Participants]
  BD | 7 | 8 | 15
  SSD | 7 | 6 | 13
Cigarettes Per Day [Mean (Standard Deviation); unit: Cigarettes] | 14.5 (3.3) | 25.2 (11) | 19.8 (9.7)
Fagerström Test for Cigarette Dependence [Mean (Standard Deviation); unit: units on a scale] — The Fagerström Test for Cigarette Dependence (FTCD) is a six-item, self-report measure of cigarette/nicotine dependence severity. Scoring on the FTCD ranges from 0 to 10. Total scores above six reflect substantial dependence severity; scores between 4- to 6 indicate moderate severity; and scores less than four reflect mild severity.
  units on a scale | 5.4 (1.6) | 6.8 (2) | 6 (1.9)
Minnesota Nicotine Withdrawal Scale [Mean (Standard Deviation); unit: units on a scale] — The Minnesota Nicotine Withdrawal Scale (MNWS) used in the present trial is a 15-item, self-report measure of tobacco withdrawal symptoms that occur when a person tries to quit smoking. Each item is scored on a 0 to 4 Likert scale (thus, 0 to 60 scoring range) with higher total scores indicating more severe tobacco withdrawal.
  units on a scale | 20.9 (12.4) | 23.5 (12.3) | 22.2 (12.2)
Questionnaire of Smoking Urges- Brief [Mean (Standard Deviation); unit: units on a scale] — The Questionnaire of Smoking Urges - Brief (QSU-B) is a 10-item self-report questionnaire that measures cravings and urges to smoke cigarettes. Each item is scored on a 1 to 7 Likert scale yielding a range of scores from 10 to 70. Higher scores registered on the QSU-B indicate more intense cravings and urges to smoke during a smoking cessation attempt.
  units on a scale | 51.1 (15) | 51.7 (15.1) | 51.4 (14.8)
Hospital Anxiety and Depression Scale (HADS) [Mean (Standard Deviation); unit: units on a scale] — The Hospital Anxiety and Depression Scale (HADS) is comprised of two separate 7-item self-report subscales with one measuring anxiety symptoms and the other measuring depressive symptoms. Each of the 7-item subscales is scored using a 0 to 3 Likert scale such that scores range from 0 to 21 units. Scores of 0 to 7 are in the normal range; 8 to 10 are borderline abnormal; and greater than 11 reflect abnormal levels of anxiety or depression.
  units on a scale
    HADS: Anxiety | 9.6 (5.9) | 12 (6.6) | 10.8 (6.3)
    HADS: Depression | 4.4 (3.9) | 6.5 (5.5) | 5.4 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Combining ACT With 2 Different Varenicline-assisted Quitting Strategies
Description: Demand for participating (# of participants recruited per month); practicality of study procedures (% participants completing study procedures); acceptability of study procedures (% participants adhering to making a quit attempt within the quit window)
Time Frame: Through completion of study, an average of 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Varenicline | Standard Dose Varenicline
Number analyzed (Participants) | 14 | 14
Participants
  Demand For Participating | 1 | 1
  Practicality of Study Procedures | 9 | 12
  Acceptability of Study Procedures | 13 | 12

2. Other Pre Specified Outcome: Nicotine Metabolite Ratio (NMR) Exploratory Aim
Description: The nicotine metabolite ratio (NMR) as measured by the ratio of 3'-hydroxycotinine (the breakdown product of cotinine) divided by the concentration of cotinine (the breakdown product of nicotine) in a smoker's serum is a biomarker of nicotine clearance. Other researchers have found that a person's NMR might influence one's response to certain smoking cessation medications. The NMR was measured in serum using electrospray ionization liquid chromatography tandem mass spectrometry technology.
Time Frame: Through completion of study, an average of 2 years
Population: Due to the small sample size and our finding that practically all smokers in this sample of persons with serious mental illness would be considered "normal metabolizers" based on population normative values, Arms/Groups were combined to maximize power and to explore whether there was any correlation between the NMR values and the incidence of adverse events. Since this was an exploratory aim, the analysis was pre-specified to include all participants regardless of varenicline condition.
Measure: Mean (Standard Deviation); unit: ratio of molar concentrations
Groups:
- Smokers With Serious Mental Illness: Participants enrolled and randomized into study
Arm/Group | Smokers With Serious Mental Illness
Number analyzed (Participants) | 28
ratio of molar concentrations | 1.20 (0.75)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the 12 week active treatment phase and for one month after treatment discontinuation (i.e. through week 16).
Arm/Group | Low Dose Varenicline | Standard Dose Varenicline
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/14
Other Adverse Events (participants affected / at risk) | 13/14 | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Varenicline (N=14) | Standard Dose Varenicline (N=14)
Depression (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Varenicline (N=14) | Standard Dose Varenicline (N=14)
Aggression (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 3 | 1
Anxiety (Psychiatric disorders) | 7 | 2
Depression (Psychiatric disorders) | 3 | 4
Panic (Psychiatric disorders) | 1 | 1
Sleep Disturbances (Psychiatric disorders) | 5 | 4
Hallucination (Psychiatric disorders) | 0 | 1
Hostility (Psychiatric disorders) | 0 | 2
Intrusive Thoughts (Psychiatric disorders) | 0 | 1
Mania (Psychiatric disorders) | 0 | 1
Paranoia (Psychiatric disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 1
Heartburn (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 1
Stomach Pain (Gastrointestinal disorders) | 1 | 1
Confusion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Fatigue (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 2
Leg Spasms (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Malaise (Nervous system disorders) | 1 | 0
Vertigo (Nervous system disorders) | 0 | 2
Confusion (General disorders) | 1 | 0
Dysgeusia (General disorders) | 7 | 6
Increased Thirst (General disorders) | 0 | 1
Increased Appetite (General disorders) | 0 | 1
Weight Gain (General disorders) | 1 | 1
Cold (Infections and infestations) | 2 | 0
Abscess (Infections and infestations) | 0 | 1
Flu (Infections and infestations) | 0 | 2
Gum Disease (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Leg Cramps (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Angina (Cardiac disorders) | 1 | 0
Increased Blood Pressure (Cardiac disorders) | 1 | 0
Coronary Heart Disease (Cardiac disorders) | 0 | 2
Palpitations (Cardiac disorders) | 1 | 0
Allergies (Immune system disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Frequent Urination (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT04011280/Prot_SAP_001.pdf